CLINICAL TRIAL: NCT00686166
Title: A Phase II Study of Oxaliplatin, Capecitabine, Cetuximab and Radiation in Pre-Operative Therapy of Rectal Cancer
Brief Title: S0713: Oxaliplatin, Capecitabine, Cetuximab, and RT Followed By Surgery in Pts W/Stage II or III Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0713; S0713 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2008-05-28; First posted 2008-05-29 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-04

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the rectum; stage IIA rectal cancer; stage IIB rectal cancer; stage IIC rectal cancer; stage IIIA rectal cancer; stage IIIB rectal cancer; stage IIIC rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Capecitabine; Oxaliplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemo + Chemo and radiation + Surgery (Experimental): Chemotherapy Cycle 1 (1 cycle is 35 days):
  * Oxaliplatin, 50 mg/m^2, IV, Days 1,8,15,22,29
  * Cetuximab, 400 mg/m^2, IV, Day 1
  * Cetuximab, 250 mg/m^2, IV, Days 8,15,22,29
  * Capecitabine, 1650 mg/m^2/day, PO, Monday-Friday (Day 1-35)
  Chemotherapy+ Radiation Cycle 2:
  * Oxaliplatin, 50 mg/m^2, IV, Days 50,57,71,78
  * Cetuximab, 250 mg/m^2, IV, Days 50,57,64,71,78
  * Capecitabine, 1650 mg/m^1, PO, Monday-Friday (Day 50-84)
  * Radiation therapy: Planning target value 1: 4500 cGy (centigray) in 25 fractions; Planning target value 2 (stage T3 patients): Boost of 540 cGy in 3 fractions; Planning target value 2 (stage T4 patients): Boost of 900 cGy in 5 fractions.
  Therapeutic Surgical procedure: Resection
  Interventions: Biological: cetuximab; Drug: capecitabine; Drug: oxaliplatin; Procedure: therapeutic surgical procedure; Radiation: radiation therapy

INTERVENTIONS:
Biological: cetuximab — Chemotherapy cycle 1: Cetuximab, 400 mg/m^2, IV, Day 1; Cetuximab, 250 mg/m^2, IV, Days 8,15,22,29
  Chemotherapy+ Radiation Cycle 2: Cetuximab, 250 mg/m^2, IV, Days 50,57,64,71,78
  Other Names: IMG-C225; Erbitux; NSC-714692
Drug: capecitabine — Chemotherapy Cycle 1: Capecitabine, 1650 mg/m^2/day, PO, Monday-Friday (Day 1-35)
  Chemotherapy+ Radiation Cycle 2: Capecitabine, 1650 mg/m^1, PO, Monday-Friday (Day 50-84)
  Other Names: Xeloda; NSC-712807
Drug: oxaliplatin — Chemotherapy Cycle 1: Oxaliplatin, 50 mg/m^2, IV, Days 1,8,15,22,29
  Chemotherapy+ Radiation Cycle 2: Oxaliplatin, 50 mg/m^2, IV, Days 50,57,71,78
  Other Names: Eloxatin; NSC-266046
Procedure: therapeutic surgical procedure — Surgical resection
  Other Names: Resection
Radiation: radiation therapy — IMRT (intensity-modulated radiation therapy)
  Other Names: RT

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying the side effects and how well giving oxaliplatin, capecitabine, and cetuximab together with radiation therapy followed by surgery works in treating patients with stage II or stage III rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the pathologic complete response rate for the combination of oxaliplatin, capecitabine, and cetuximab alone and concurrently with external beam radiotherapy for patients with adenocarcinoma of the rectum, stages II and III with wild-type K-ras.
* To estimate the 3-year disease-free survival probability in this patient population when treated with this regimen.
* To assess the frequency and severity of toxicities associated with this regimen in these patients.
* To explore, preliminarily, the association between expression levels of genes involved in the DNA repair, EGFR (epidermal growth factor receptor), angiogenesis, and 5-FU pathway (i.e., k-ras, TS [Thymidylate Synthase], ERCC-1 [excision repair cross complementing-1), TP [Thymidine phosphorylase], DPD [Dihydropyrimidine dehydrogenase], EGFR, VEGF [vascular endothelial growth factor], and IL-8 [interleukin-8]) and pathologic complete response. (Due to advances in methodology, the translational medicine objectives are being reconsidered. Therefore, results for this objective are not reported)
* To explore, preliminarily, the intratumoral gene expression levels of these genes after completion of study treatment.(Due to advances in methodology, the translational medicine objectives are being reconsidered. Therefore, results for this objective are not reported)
* To obtain, preliminarily, data on genomic polymorphisms of these genes for correlation with clinical outcome and toxicity. (Due to advances in methodology, the translational medicine objectives are being reconsidered. Therefore, results for this objective are not reported)

OUTLINE: This is a multicenter study.

* Neoadjuvant therapy (course 1): Patients receive oxaliplatin IV over 2 hours once a week for 5 weeks, oral capecitabine twice daily 5 days a week for 5 weeks, and cetuximab IV over 1-2 hours once a week for 5 weeks.
* Neoadjuvant therapy with concurrent radiotherapy (course 2): Beginning two weeks later, patients receive oxaliplatin IV over 2 hours once a week in weeks 1, 2, 4, and 5. Patients also receive capecitabine and cetuximab as in course 1. Patients also undergo external beam radiotherapy 5 days a week for 5 weeks beginning in week 1.

Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo surgery 3-8 weeks after completion of chemoradiotherapy.

Blood samples are collected for germline polymorphism testing and tissue samples are collected and assessed for gene expression analysis.

After completion of study treatment, patients are followed every 6 months for 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven primary adenocarcinoma of the rectum

  * Stage II or III disease
  * The distal border of the tumor must be at or below the peritoneal reflection, defined as within 12 cm of the anal verge by proctoscopic examination
  * No recurrent disease
* Must have wild-type k-ras status
* Measurable and/or nonmeasurable disease

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Leukocyte count ≥ 3,000/mcL
* Granulocyte count ≥ 1,500/mcL
* Platelet count ≥ 100,000/mcL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* SGOT (serum glutamate oxaloacetate transaminase) or SGPT (serum glutamate pyruvate transaminase)≤ 2.5 times ULN
* Creatinine clearance > 50 mL/min
* No prior severe reaction to a monoclonal antibody
* Willing to have specimens submitted
* No peripheral neuropathy ≥ grade 2
* No known existing uncontrolled coagulopathy
* No evidence of current high-grade obstruction

  * At least 2 weeks since prior diverting procedure
* No history of allergy to platinum compounds or to antiemetics appropriate for administration in conjunction with protocol treatment
* No prior unanticipated severe reaction to fluoropyrimidine therapy or known sensitivity to fluorouracil or known DPD deficiency
* No active inflammatory bowel disease, malabsorption syndrome, or inability to swallow that would impair the ingestion or absorption of capecitabine
* No uncontrolled intercurrent illness
* No ongoing or active infection
* No symptomatic congestive heart failure or unstable angina pectoris
* No cardiac arrhythmia or myocardial infarction within the past 12 months
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No prior malignancy allowed except for adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or other cancer from which the patient has been disease-free for 5 years

PRIOR CONCURRENT THERAPY:

* Recovered from any recent major surgeries (e.g., coronary artery bypass graft, transurethral resection of prostate, or abdominal surgery)
* No prior chemotherapy, radiotherapy, or targeted therapy for this tumor
* More than 4 weeks since prior investigational agents
* No concurrent anti-retroviral therapy for HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2009-02; Primary Completion 2014-07 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia G. Leichman, MD, Study Chair — Breastlink
Locations (130):
- United States (130):
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Arizona Cancer Center at UMC Orange Grove, Tucson, Arizona
  - Arizona Cancer Center at University Medical Center North, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Sutter Health - Western Division Cancer Research Group, Novato, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Sutter Cancer Center at Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Sutter Solano Medical Center, Vallejo, California
  - Memorial Hospital Cancer Center - Colorado Springs, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Hays Medical Center, Hays, Kansas
  - Hutchinson Hospital Corporation, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Kansas City Cancer Centers - West, Kansas City, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Mount Carmel Regional Cancer Center, Pittsburg, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Kansas City Cancer Center - Shawnee Mission, Shawnee Mission, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Kansas City Cancer Centers - South, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Kansas City Cancer Centers - East, Lee's Summit, Missouri
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - AnMed Cancer Center, Anderson, South Carolina
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - U.T. Medical Center Cancer Institute, Knoxville, Tennessee
  - Southwest Regional Cancer Center - Central, Austin, Texas
  - Texas Oncology, PA at Texas Oncology Cancer Center - Central, Austin, Texas
  - Texas Oncology, PA at South Austin Cancer Center, Austin, Texas
  - Texas Oncology, PA - Austin North, Austin, Texas
  - Texas Oncology, PA - Cedar Park, Cedar Park, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - St. Luke's Texas Cancer Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - Texas Oncology, PA - Seton Williamson, Round Rock, Texas
  - Texas Oncology, PA at Texas Cancer Center Round Rock, Round Rock, Texas
  - Texas Oncology, PA - San Marcos, San Marcos, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Island Hospital Cancer Care Center at Island Hospital, Anacortes, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Highline Medical Center Cancer Center, Burien, Washington
  - Swedish Medical Center - Issaquah Campus, Issaquah, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemo + Chemo and Radiation + Surgery
Started | 83
Eligible | 78
Eligible and Began Protocol Therapy | 74
Completed | 63
Not Completed | 20
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 1
Not completed — Progression/Relapse | 1
Not completed — Death | 1
Not completed — Not Protocol Specified | 1
Not completed — Ineligible | 5
Not completed — Did not begin protocol therapy | 4

BASELINE CHARACTERISTICS:
Population: Eligible patients who began protocol therapy.
Arm/Group | Chemo + Chemo and Radiation + Surgery
Number analyzed (Participants) | 74
Age, Continuous [Median (Full Range); unit: years] | 56.4 [25.5 to 77.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 63
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate
Description: Pathologic response is evaluated after the patient has had surgery, and is based on local pathology review of the resected surgical specimen, according to the following: a) Pathologic complete response (pCR): on review of the resected rectal specimen and accompanying lymph nodes, no cancer is recognized by the pathologist; b) Microscopic cancer: gross tumor is not seen by the pathologist but tumor remains in the microscopic analysis of any part of the entire specimen; c) no response: gross cancer is found on pathologic examination of the resected rectal cancer and draining lymph nodes.
Time Frame: 15-20 weeks from registration
Population: Eligible and analyzable patients with available data. It was assumed that a pathologic complete response was not achieved for patients who do not receive surgery or for whom a surgical specimen is lacking. These patients were included in the denominator.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemo + Chemo and Radiation + Surgery
Number analyzed (Participants) | 72
percentage of participants | 25 [16 to 37]
Statistical Analysis 1: Comparison: Chemo + Chemo and Radiation + Surgery; Test type: Superiority or Other; p = 0.18, Exact binomal test

2. Secondary Outcome: 3-year Disease-free Survival
Description: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression free are censored at date of last contact.
Time Frame: 3 years
Population: Eligible and analyzable patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemo + Chemo and Radiation + Surgery
Number analyzed (Participants) | 74
percentage of participants | 68 [57 to 78]

3. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to This Regimen.
Description: Only adverse events that are possibly, probably or definitely related to study regimen are reported.
Time Frame: Up to 4 years
Population: Eligible patients who received any treatment and were assessed for adverse events are included in this summary.
Measure: Number; unit: Participants
Groups:
- Chemotherapy: Patients receive oxaliplatin 50 mg/m^2 IV (Days 1, 8, 15, 22, 29), cetuximab 400 mg/m^2 IV (Day 1), cetuximab 250 mg/m^2 IV (Days 8, 15, 22, 29), capecitabine 1650 mg/m^2 PO (Monday-Friday, Day 1-35). Cycle is 35 days, followed by a 14-day break.
- Chemotherapy + Radiation: Patients receive oxaliplatin 50 mg/m^2 IV (Days 50, 57, 71, 78), cetuximab 250 mg/m^2 IV (Days 50, 57, 64, 71, 78), capecitabine 1650 mg/m^2 PO (Monday-Friday, Day 50-84). Radiation therapy begins on Day 50. Dose and length of treatment are dependent on technique used and clinical stage. Planned target value 1: 4500 cGy (centigray) in 25 fractions; Planned target value 2 (stage 3 patients): Boost of 540 cGy in 3 fractions; Planning target value 2 (stage T4 patients): Boost of 900 cGy in 5 fractions.
- Tumor Resection: Surgery must take place between 3 - 8 weeks after completion of chemoradiation. Surgical resections should adhere to the principles of total mesorectal excision as described by Heald.
Arm/Group | Chemotherapy | Chemotherapy + Radiation | Tumor Resection
Number analyzed (Participants) | 74 | 68 | 63
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 15 | 11 | 3
  AST, SGOT | 15 | 12 | 2
  Acidosis (metabolic or respiratory) | 1 | 0 | 0
  Adult respiratory distress syndrome (ARDS) | 1 | 0 | 0
  Albumin, serum-low (hypoalbuminemia) | 11 | 10 | 7
  Alkaline phosphatase | 4 | 5 | 3
  Allergic reaction/hypersensitivity | 0 | 1 | 0
  Allergic rhinitis | 2 | 1 | 0
  Amylase | 0 | 0 | 1
  Anorexia | 20 | 18 | 9
  Bicarbonate, serum-low | 1 | 1 | 2
  Bilirubin (hyperbilirubinemia) | 5 | 3 | 2
  Blood/Bone Marrow-Other | 2 | 1 | 1
  Bone: spine-scoliosis | 1 | 0 | 0
  Bruising (in absence of Gr 3-4 thrombocytopenia) | 0 | 1 | 0
  Burn | 0 | 2 | 0
  Calcium, serum-low (hypocalcemia) | 8 | 13 | 9
  Coagulation-Other | 1 | 0 | 0
  Colitis | 1 | 0 | 0
  Confusion | 2 | 0 | 0
  Constipation | 34 | 24 | 5
  Constitutional Symptoms-Other | 2 | 1 | 0
  Cough | 2 | 6 | 1
  Creatinine | 2 | 0 | 4
  Cystitis | 0 | 0 | 1
  Cytokine release syndrome/acute infusion reaction | 1 | 1 | 0
  Dehydration | 8 | 11 | 1
  Dermatology/Skin-Other | 1 | 2 | 0
  Diarrhea | 34 | 48 | 10
  Distention/bloating, abdominal | 0 | 1 | 0
  Dizziness | 10 | 7 | 1
  Dry mouth/salivary gland (xerostomia) | 7 | 6 | 0
  Dry skin | 20 | 16 | 2
  Dysphagia (difficulty swallowing) | 2 | 1 | 0
  Dyspnea (shortness of breath) | 5 | 4 | 1
  Edema: limb | 1 | 1 | 2
  Enteritis (inflammation of the small bowel) | 1 | 2 | 0
  Extrapyramidal/involuntary movement/restlessness | 1 | 0 | 1
  Fatigue (asthenia, lethargy, malaise) | 48 | 41 | 22
  Fever in absence of neutropenia, ANC lt1.0x10e9/L | 4 | 4 | 2
  Flatulence | 0 | 5 | 0
  Flu-like syndrome | 0 | 1 | 0
  Flushing | 2 | 0 | 0
  Gastritis (including bile reflux gastritis) | 2 | 1 | 1
  Gastrointestinal-Other | 2 | 6 | 1
  Glucose, serum-high (hyperglycemia) | 13 | 12 | 6
  Hair loss/Alopecia (scalp or body) | 4 | 3 | 0
  Heartburn/dyspepsia | 13 | 4 | 0
  Hemoglobin | 13 | 19 | 21
  Hemolysis | 1 | 1 | 0
  Hemorrhage, GI - Rectum | 9 | 6 | 3
  Hemorrhage/Bleeding-Other | 0 | 2 | 0
  Hemorrhage/bleeding w/surgery, intra- or post-op | 0 | 0 | 2
  Hemorrhoids | 0 | 5 | 1
  Hepatobiliary/Pancreas-Other | 1 | 0 | 0
  Hiccoughs (hiccups, singultus) | 2 | 1 | 2
  Hot flashes/flushes | 0 | 1 | 0
  Hyperpigmentation | 0 | 5 | 1
  Hypertension | 3 | 2 | 1
  Hypotension | 4 | 2 | 0
  INR (of prothrombin time) | 0 | 1 | 1
  Ileus, GI (functional obstruction of bowel) | 0 | 0 | 1
  Incontinence, anal | 1 | 4 | 0
  Incontinence, urinary | 1 | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - UTI | 2 | 1 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Vagina | 0 | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Wound | 0 | 0 | 1
  Infection with unknown ANC - Abdomen NOS | 0 | 0 | 2
  Infection with unknown ANC - Anal/perianal | 0 | 0 | 1
  Infection with unknown ANC - Sinus | 1 | 0 | 0
  Infection with unknown ANC - Urinary tract NOS | 1 | 0 | 0
  Infection-Other | 0 | 1 | 1
  Injection site reaction/extravasation changes | 1 | 0 | 0
  Insomnia | 4 | 6 | 1
  Irregular menses (change from baseline) | 0 | 1 | 0
  Leak (including anastomotic), GU - Stoma | 0 | 0 | 1
  Leukocytes (total WBC) | 2 | 6 | 3
  Lipase | 1 | 0 | 1
  Lymphatics-Other | 0 | 1 | 0
  Lymphopenia | 4 | 13 | 9
  Magnesium, serum-high (hypermagnesemia) | 2 | 0 | 0
  Magnesium, serum-low (hypomagnesemia) | 3 | 4 | 2
  Metabolic/Laboratory-Other | 3 | 4 | 2
  Mood alteration - agitation | 1 | 0 | 0
  Mood alteration - anxiety | 6 | 3 | 1
  Mood alteration - depression | 4 | 2 | 0
  Mucositis/stomatitis (clinical exam) - Anus | 0 | 1 | 0
  Mucositis/stomatitis (clinical exam) - Oral cavity | 14 | 4 | 0
  Mucositis/stomatitis (functional/symp) - Anus | 1 | 1 | 0
  Mucositis/stomatitis (functional/symp) - Oral cav | 9 | 2 | 0
  Mucositis/stomatitis (functional/symp) - Rectum | 0 | 4 | 0
  Muscle weakness, not d/t neuropathy - Extrem-lower | 3 | 2 | 0
  Muscle weakness, not d/t neuropathy - Extrem-upper | 1 | 0 | 0
  Muscle weakness, not d/t neuropathy - body/general | 3 | 4 | 1
  Musculoskeletal/Soft Tissue-Other | 0 | 1 | 0
  Nail changes | 2 | 3 | 1
  Nasal cavity/paranasal sinus reactions | 0 | 1 | 0
  Nausea | 37 | 25 | 7
  Neurology-Other | 2 | 0 | 0
  Neuropathy: motor | 0 | 1 | 0
  Neuropathy: sensory | 38 | 34 | 17
  Neutrophils/granulocytes (ANC/AGC) | 4 | 9 | 2
  Obstruction, GI - Rectum | 1 | 1 | 0
  Obstruction, GI - Small bowel NOS | 3 | 0 | 0
  Ocular/Visual-Other | 1 | 0 | 0
  PTT (Partial thromboplastin time) | 0 | 0 | 1
  Pain - Abdomen NOS | 8 | 19 | 7
  Pain - Anus | 0 | 5 | 1
  Pain - Back | 4 | 1 | 1
  Pain - Bone | 0 | 1 | 0
  Pain - Chest/thorax NOS | 1 | 0 | 0
  Pain - Esophagus | 0 | 1 | 0
  Pain - Extremity-limb | 3 | 4 | 1
  Pain - Face | 1 | 0 | 0
  Pain - Head/headache | 10 | 3 | 0
  Pain - Joint | 5 | 2 | 1
  Pain - Kidney | 1 | 0 | 0
  Pain - Muscle | 1 | 2 | 1
  Pain - Oral cavity | 2 | 0 | 0
  Pain - Pelvis | 1 | 1 | 1
  Pain - Perineum | 0 | 1 | 1
  Pain - Rectum | 5 | 20 | 17
  Pain - Urethra | 0 | 1 | 1
  Pain - Vagina | 0 | 2 | 0
  Pain-Other | 2 | 3 | 0
  Phlebitis (including superficial thrombosis) | 1 | 0 | 0
  Phosphate, serum-low (hypophosphatemia) | 1 | 0 | 0
  Photosensitivity | 2 | 1 | 0
  Platelets | 9 | 13 | 6
  Pleural effusion (non-malignant) | 0 | 1 | 0
  Potassium, serum-high (hyperkalemia) | 2 | 0 | 1
  Potassium, serum-low (hypokalemia) | 14 | 14 | 4
  Proctitis | 0 | 5 | 1
  Pruritus/itching | 15 | 5 | 0
  Pulmonary hypertension | 1 | 0 | 0
  Pulmonary/Upper Respiratory-Other | 0 | 2 | 0
  Rash/desquamation | 7 | 5 | 3
  Rash: acne/acneiform | 64 | 42 | 9
  Rash: dermatitis associated w/Chemoradiation | 0 | 7 | 1
  Rash: dermatitis associated w/radiation | 0 | 4 | 2
  Rash: erythema multiforme | 0 | 2 | 0
  Rash: hand-foot skin reaction | 12 | 12 | 4
  Renal failure | 1 | 0 | 0
  Renal/Genitourinary-Other | 2 | 0 | 1
  Rigors/chills | 3 | 1 | 2
  SVT and nodal arrhythmia - Atrial fibrillation | 1 | 0 | 0
  SVT and nodal arrhythmia - Atrial tachycardia/PAT | 0 | 0 | 1
  SVT and nodal arrhythmia - Sinus tachycardia | 3 | 0 | 1
  Sexual/Reproductive Function-Other | 1 | 0 | 0
  Sodium, serum-high (hypernatremia) | 2 | 0 | 0
  Sodium, serum-low (hyponatremia) | 7 | 6 | 6
  Somnolence/depressed level of consciousness | 0 | 2 | 0
  Sweating (diaphoresis) | 1 | 0 | 0
  Syncope (fainting) | 0 | 0 | 1
  Taste alteration (dysgeusia) | 3 | 4 | 1
  Thrombosis/embolism (vascular access-related) | 1 | 0 | 0
  Thrombosis/thrombus/embolism | 1 | 0 | 0
  Tinnitus | 0 | 1 | 0
  Tremor | 1 | 0 | 0
  Urinary frequency/urgency | 0 | 4 | 1
  Urinary retention (including neurogenic bladder) | 0 | 2 | 6
  Vascular-Other | 1 | 0 | 0
  Ventricular arrhythmia - Ventricular tachycardia | 0 | 1 | 0
  Vision-blurred vision | 1 | 0 | 0
  Vomiting | 13 | 5 | 4
  Weight gain | 0 | 1 | 0
  Weight loss | 11 | 15 | 12
  Wound complication, non-infectious | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: Eligible patients who received any treatment and were assessed for adverse events are included in the adverse event summaries.
Arm/Group | Chemotherapy | Chemotherapy + Radiation | Tumor Resection
Serious Adverse Events (participants affected / at risk) | 1/74 | 0/68 | 0/63
Other Adverse Events (participants affected / at risk) | 73/74 | 66/68 | 51/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (N=74) | Chemotherapy + Radiation (N=68) | Tumor Resection (N=63)
Death - Multi-organ failure (General disorders) | 1 | 0 | 0
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 | 0 | 0
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (N=74) | Chemotherapy + Radiation (N=68) | Tumor Resection (N=63)
Hemoglobin (Blood and lymphatic system disorders) | 13 | 19 | 21
Constipation (Gastrointestinal disorders) | 34 | 24 | 5
Diarrhea (Gastrointestinal disorders) | 34 | 48 | 10
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 7 | 6 | 0
Flatulence (Gastrointestinal disorders) | 0 | 5 | 0
Gastrointestinal-Other (Gastrointestinal disorders) | 2 | 6 | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 13 | 4 | 0
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 9 | 6 | 3
Hemorrhoids (Gastrointestinal disorders) | 0 | 5 | 1
Incontinence, anal (Gastrointestinal disorders) | 1 | 4 | 0
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 14 | 4 | 0
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 9 | 2 | 0
Mucositis/stomatitis (functional/symp) - Rectum (Gastrointestinal disorders) | 0 | 4 | 0
Nausea (Gastrointestinal disorders) | 37 | 25 | 7
Pain - Abdomen NOS (Gastrointestinal disorders) | 8 | 19 | 7
Pain - Anus (Gastrointestinal disorders) | 0 | 5 | 1
Pain - Rectum (Gastrointestinal disorders) | 5 | 20 | 17
Proctitis (Gastrointestinal disorders) | 0 | 5 | 1
Vomiting (Gastrointestinal disorders) | 13 | 5 | 4
Fatigue (asthenia, lethargy, malaise) (General disorders) | 48 | 41 | 22
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 4 | 4 | 2
Rash: dermatitis associated w/Chemoradiation (Injury, poisoning and procedural complications) | 0 | 7 | 1
Rash: dermatitis associated w/radiation (Injury, poisoning and procedural complications) | 0 | 4 | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 15 | 11 | 3
AST, SGOT (Investigations) | 15 | 12 | 2
Alkaline phosphatase (Investigations) | 4 | 5 | 3
Bilirubin (hyperbilirubinemia) (Investigations) | 5 | 3 | 2
Creatinine (Investigations) | 2 | 0 | 4
Leukocytes (total WBC) (Investigations) | 2 | 6 | 3
Lymphopenia (Investigations) | 4 | 13 | 9
Metabolic/Laboratory-Other (Investigations) | 3 | 4 | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 4 | 9 | 2
Platelets (Investigations) | 9 | 13 | 6
Weight loss (Investigations) | 11 | 15 | 12
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 11 | 10 | 7
Anorexia (Metabolism and nutrition disorders) | 20 | 18 | 9
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 8 | 13 | 9
Dehydration (Metabolism and nutrition disorders) | 8 | 11 | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 13 | 12 | 6
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3 | 4 | 2
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 14 | 14 | 4
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 7 | 6 | 6
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 3 | 4 | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 3 | 4 | 1
Pain - Joint (Musculoskeletal and connective tissue disorders) | 5 | 2 | 1
Dizziness (Nervous system disorders) | 10 | 7 | 1
Neuropathy: sensory (Nervous system disorders) | 38 | 34 | 17
Pain - Head/headache (Nervous system disorders) | 10 | 3 | 0
Taste alteration (dysgeusia) (Nervous system disorders) | 3 | 4 | 1
Insomnia (Psychiatric disorders) | 4 | 6 | 1
Mood alteration - anxiety (Psychiatric disorders) | 6 | 3 | 1
Mood alteration - depression (Psychiatric disorders) | 4 | 2 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 4 | 1
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 0 | 2 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 20 | 16 | 2
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4 | 3 | 0
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 5 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 15 | 5 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 | 5 | 3
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 64 | 42 | 9
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 12 | 12 | 4
Hypotension (Vascular disorders) | 4 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No